CLINICAL TRIAL: NCT02184104
Title: Pharmacokinetics and Pharmacodynamics of a 100 mg Caffeine Dose After Oral Consumption of an Energy Drink or Inhalation Using the Aeroshot Administration Device
Brief Title: Caffeine Disposition After Inhalation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13-02648-FB; 1R03DA035347-01A1 (NIH)
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: caffeine; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aeroshot (Active Comparator): A single 100 mg caffeine dose administered using the Aeroshot device.
  Interventions: Dietary Supplement: Caffeine
- Energy Drink (Active Comparator): A single 100 mg caffeine dose administered as an oral solution.
  Interventions: Dietary Supplement: Caffeine

INTERVENTIONS:
Dietary Supplement: Caffeine

SUMMARY:
The purpose of this study is to determine how fast caffeine gets into your body with a product called Aeroshot™. Aeroshot™ is a lipstick sized device that you slide open and then put your mouth over the opening and inhale. A fine powder containing 100 mg of caffeine is deposited on your tongue and the inside of your mouth. Caffeine will be absorbed through the membranes in your mouth or swallowed and then absorbed in your stomach. We will compare the absorption of caffeine after using the Aeroshot™ with the absorption after drinking an energy drink by taking 15 blood samples over 8 hours and measuring the caffeine levels in your blood. You will also be asked to fill out some scales to measure the effects you feel after the caffeine dose. We hypothesize that caffeine absorption after inhalation will be faster than after an energy drink.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* non-smoker

Exclusion Criteria:

* Take chronic medication
* Co-existing diseases
* Platelet count less than 100,000/uL (per microliter)
* Acute or chronic psychiatric condition
* Consume more than 300 mg of caffeine per day
* Participated in another study within last 30 days or donated blood in last 6 weeks

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Caffeine plasma concentration | 0, 1, 2, 5, 10, 15, 20, 30, 40, 60 minutes and 2, 3, 4, 6, 8 hours
  These are the collection times of blood samples relative to when the caffeine dose was consumed.

SECONDARY OUTCOMES:
Caffeine effects | 0, 1, 2, 5, 10, 15, 20, 30, 40, 60 minutes, and 2, 3, 4, 6, 8 hours
  Subjects will complete seven analog scales to assess the effects that they feel after the caffeine dose.

OTHER OUTCOMES:
Cardiovascular effects | 0, 1, 2, 5, 10, 15, 20, 30, 40, 60 minutes, and 2, 3, 4, 6, 8 hours
  The heart rate and blood pressure will be recorded at the time of each blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Laizure, Pharm.D., Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No